CLINICAL TRIAL: NCT02744430
Title: A Double Blind Placebo Control Trial of Mirabegron for Medical Expulsive Therapy and to Manage Stent Pain for Ureteral Stones(Protocol # 01-16-20-02)
Brief Title: Mirabegron as Medical Expulsive Therapy (MET) for Ureteral Stones and Ureteral Stent Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Wesley Adam Mayer, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-38959
Record Dates: First submitted 2016-04-12; First posted 2016-04-20 (Estimated); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Ureteral Obstruction; Flank Pain
Keywords: Medical expulsive therapy; ureteral stone; stent pain
MeSH Terms: conditions — Ureteral Obstruction; Flank Pain; Ureterolithiasis | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Active (Active Comparator): Mirabegron 50 mg orally once every 24 hours starting immediately
  Interventions: Drug: Mirabegron
- Arm 2 - Placebo (Placebo Comparator): Placebo orally once every 24 hours starting immediately
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mirabegron — Randomized 1:1 ratio using a randomized block design, stratified by stone size (≤5 mm versus >5 mm) and location (upper versus lower ureter). The randomization will be implemented through a database with software designed by the Director of Research Informatics at the Baylor College of Medicine's Dan Duncan Institute of Clinical and Translational Research. It will be a HIPPA-compliant secure database accessible via internet.
  Other Names: Myrbetriq
  Arms: Arm 1 - Active
Other: Placebo — Randomized 1:1 ratio using a randomized block design, stratified by stone size (≤5 mm versus >5 mm) and location (upper versus lower ureter). The randomization will be implemented through a database with software designed by the Director of Research Informatics at the Baylor College of Medicine's Dan Duncan Institute of Clinical and Translational Research. It will be a HIPPA-compliant secure database accessible via internet.
  Arms: Arm 2 - Placebo

SUMMARY:
The study will be a prospective randomized double-blind placebo-controlled trial of mirabegron for medical expulsive therapy (MET) in patients with a CT (Computed Tomography) scan-proven ureteral stone between 4 to 10 mm undergoing expectant management.

DETAILED DESCRIPTION:
The study will be a prospective randomized double-blind placebo-controlled trial of mirabegron for medical expulsive therapy (MET) in patients with a CT scan-proven ureteral stone between 4 to 10 mm undergoing expectant management. Subjects will be distributed at a 1:1 ratio between the control and treatment groups. The treatment group will receive mirabegron and the control groups will receive a placebo. Both groups will receive analgesics and hydration will be recommended. All subjects will then be followed for 30 days to determine the proportion of subjects with spontaneous passage. Patients will record narcotic usage and pain scores during this time. If there is stone persistence in the ureter based on imaging (CT scan of the abdomen and pelvis versus renal ultrasound plus KUB), then the patient will undergo ureteroscopy with stent placement. In these patients, treatment will continue while the stent is in place and patients will fill out a validated questionnaire regarding stent pain.

ELIGIBILITY:
Inclusion Criteria:

* Single unilateral ureteral calculus 4 to 10 mm visible on CT scan within the ureter
* Serum creatinine within normal range
* Ability to tolerate oral fluids and oral pain medication
* Able to make informed medical decisions regarding consent
* Willingness to follow-up in the Urology Clinic in approximately 30 day
* Willing to undergo ureteroscopic extraction should the stone not pass in this time period

Exclusion Criteria:

* Adults unable to consent
* Age less than 18
* Multiple stones
* Solitary kidney
* Horseshoe kidney
* On immunosuppressant therapy
* On digoxin
* Uncontrolled hypertension (Systolic blood pressure > 170, diastolic blood pressure > 110)
* History of ureteral surgery or previous endoscopic procedure
* Allergy to mirabegron
* Current calcium antagonist or corticosteroid or tamsulosin usage
* Patients already taking a beta-adrenergic agonist medication
* Renal insufficiency [Glomerular Filtration Rate (GFR) less than 60]
* Patients with Childs B and C liver failure
* Signs of infection i. Temperature greater than 38 degrees Celsius ii. Urinalysis with any of the following positive:

  1. Positive nitrites
  2. White blood cell count greater than 15/hpf (high powered field)
  3. Positive urine culture [defined as a single isolated bacterial species population of greater than 100,000 Colony Forming Units (CFU)]
* Patients with chronic pain already undergoing treatment with narcotic medications
* Pregnant women and nursing mothers
* Prisoners
* No working phone number

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-22 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley A. Mayer, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be published in a aggregate format after completion of study.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Arm 1 - Active | Arm 2 - Placebo
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Active | Arm 2 - Placebo | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.0) | 40.8 (9.1) | 40.45 (20.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 14 | 10 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 1 | 1 | 2
  Black/African | 1 | 0 | 1
  White | 16 | 16 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 16 | 33
CBC WBC [Mean (Standard Deviation); unit: 10^9 cells/L] | 10.7 (2.5) | 11.1 (2.6) | 10.9 (5.1)
CBC Hgb [Mean (Standard Deviation); unit: grams/dL] | 10.7 (2.5) | 11.1 (2.6) | 10.9 (5.1)
CBC Platelets [Mean (Standard Deviation); unit: "10^10 platelets per liter] | 15.1 (1.6) | 13.6 (1.3) | 14.35 (2.9)
BMP Creatinine [Mean (Standard Deviation); unit: mg/dl] | 1 (0.2) | .9 (0.2) | 0.95 (.4)
BMP Potassium [Mean (Standard Deviation); unit: mmol/L] | 4 (0.4) | 3.8 (0.4) | 3.9 (.8)
BMP Calcium [Mean (Standard Deviation); unit: mmol/L] | 1.1 (.1) | 1.2 (0.1) | 1.15 (.2)
Stone Size [Mean (Standard Deviation); unit: mm] | 5.5 (1.5) | 5.4 (1.6) | 5.45 (3.1)
UA RBC [Mean (Standard Deviation); unit: RBC/HPF] | 20 (4.0) | 19 (5.0) | 19.5 (11.0)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 14 | 10 | 24
Previous Stone [Number; unit: count of participants]
  Yes | 6 | 11 | 8.5
  No | 11 | 5 | 8
Stone Location [Count of Participants; unit: Participants]
  Upper | 3 | 11 | 14
  Lower | 14 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Stone Passage Using Fisher's Exact Test
Description: The primary outcome was stone passage rate at 30-days defined by either imaging (CT or Renal Ultrasound/KUB) or identification of stone using a straining device.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Active | Arm 2 - Placebo
Number analyzed (Participants) | 17 | 16
Participants | 8 | 5

2. Secondary Outcome: Comparison of Pain Levels Between Treatment Groups Using the Wong-Baker Pain Rating Scale
Description: Pain measures between treatment groups will be measured daily for each patient by using the Wong-Baker Pain Rating Scale. The Questionnaire will be observed in patients who require surgical intervention, and will be observed during study visit. A general linear model will be used to compare Wong-Baker pain scores between the treated and placebo groups. The model will also be used to explore associations between pain scores and demographic or clinical characteristics adjusting for treatment group.
Time Frame: 2 months
Population: Comparisons between arms were calculated with ttest, Wilcoxon rank sum, and Fisher's exact test. Regression assessed odds of stone passageby 30 day visit by treatment arm. Time-to-stone pass was analyzed using Kaplan-Meier curves, log rank test,Cox proportional hazards regression. Patients who didn't pass stone were censored at last follow-up date. Wong-Baker Pain Rating Scale has zero to ten range. Zero represents no pain and ten represents worst.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Arm 1 - Active | Arm 2 - Placebo
Number analyzed (Participants) | 17 | 16
units on a scale | 0.21 [0 to 10] | 0.19 [0 to 10]

ADVERSE EVENTS:
Time Frame: The research study staff will contact the subject by phone approximately 7, 21 and 30 days after Visit 1. Research staff will assess ureteral pain, medication/strainer compliance, and adverse events. Next
Description: Safety outcomes will be reported when they happened. Suspected serious adverse events will be graded at site by the principal investigator. Safety events will be monitored by Astellas research ethics committee, and MHRA.
  Reporting of unanticipated problems will be in accordance to the current IRB guidelines and FDA regulations.
Arm/Group | Arm 2 - Placebo | Arm 1 - Active
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Consent form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT02744430/Prot_SAP_ICF_002.pdf
  • Informed Consent Form: Consent Form (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT02744430/ICF_003.pdf